CLINICAL TRIAL: NCT05417230
Title: RC48-ADC in Combination With Envolizumab for the First-line Treatment of Locally Advanced or Metastatic Biliary Tract Cancer With Positive HER-2: A Prospective, Single-arm Phase II Trial.
Brief Title: RC48-ADC Combinatioed Envolizumab in Locally Advanced or Metastatic Biliary Tract Cancer With Positive HER-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Liangjun Zhu M.M., chief physician, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-030
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — envafolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC plus envafolimab (Experimental)
  Interventions: Drug: RC48-ADC; Drug: Envafolimab

INTERVENTIONS:
Drug: RC48-ADC — 2.5mg/kg, IV, d1, every 2 weeks;
Drug: Envafolimab — 200mg, SC, d1, every 2 weeks;

SUMMARY:
This study was a prospective, single-arm phase II clinical trial to observe and evaluate the efficacy and safety of RC48-ADC combined envafolimab in the first-line treatment of locally advanced or metastatic biliary tract cancer with positive HER-2.

ELIGIBILITY:
Inclusion Criteria:

* 18 years;

  * ECOG 0-1;
  * patients diagnosed by pathological or cytological diagnosis of locally advanced or metastatic biliary tract cancer (include intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, gallbladder and ampullary carcinoma);
  * life expectancy of at least 3 months;
  * HER2 IHC 2+ or 3+;
  * At least one measurable objective tumor lesion according to RECIST 1.1;
  * Not received systemic chemotherapy in the past. Patients who have completed adjuvant therapy or neoadjuvant therapy before the start of the chemotherapy regimen in this trial 6 months ago can be included in this trial.
  * satisfactory main organ function (laboratory test must meet the following criteria): hemoglobin (HGB) ≥90g/L, neutrophil count (ANC) ≥1.5×109/L, platelet count (PLT) ≥80×109/L, Serum creatinine (CR) ≤1.5 upper normal limitation (UNL), total bilirubin (TBil) ≤1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 UNL (For patients with liver metastasis, the AST/ALT must be ≤5.0 UNL), left ventricular ejection fraction (LVEF) ≥ 50%;
  * Subjects of childbearing potential must use an appropriate method of contraception during the study period and within 120 days after the end of the study, have a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating subjects;

Exclusion Criteria:

* Previously received drug therapy against PD-1/PD-L1 inhibitor and other Antibody conjugate drug (Such as T-DM1 and DS8201);
* Allergic to the active ingredients or excipients of the study drug;
* biliary obstruction were excluded. Unless blockage is treated locally, such as endoscopic stenting, percutaneous hepatic drainage, etc., total bilirubin is reduced below the upper limit of 1.5 UNL;
* A history of malignancies other than biliary tract malignancies (other than cured carcinoma in situ of the cervix or basal cell carcinoma of the skin and other malignancies cured for 5 years);
* Received major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of study treatment; or had a long-term unhealed wound or fracture;
* Unsuitable for the study or other chemotherapy determined by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  Objective response rate

SECONDARY OUTCOMES:
DCR | 9 months
  Disease Control Rate
DOR | 12 months
  Duration of Response
PFS | 6 months
  Progression Free Survival
OS | 12 months
  Overall Survival
AEs | 12 months
  Percentage of participants experiencing grade 3-5 adverse events

OTHER OUTCOMES:
ctDNA | 12 months
  circulating tumor DNA

CONTACTS AND LOCATIONS:
Overall Officials: Liangjun Zhu, Study Chair — Jiangsu Cancer Institute & Hospital

IPD SHARING:
Plan to Share IPD: No